CLINICAL TRIAL: NCT07274878
Title: Simple Interrupted Skin Sutures Versus Subcuticular Suture Plus Subcutaneous Drain for Wound Outcomes After Open Appendectomy
Brief Title: Interrupted vs Subcuticular Sutures With Drain in Open Appendectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Rajab Abdulwahab Abdulwahab, Docter, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IVSSDOART
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sutures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subcuticular suture plus subcutaneous drain (Experimental)
  Interventions: Procedure: subcuticular suture plus subcutaneous drain

INTERVENTIONS:
Procedure: subcuticular suture plus subcutaneous drain — Subcuticular suture plus subcutaneous drain uses a continuous absorbable subcuticular stitch combined with a drain placed in the subcutaneous layer to reduce dead space and fluid collection-offering both cosmetic closure and added infection-prevention compared with standard skin-only techniques.

SUMMARY:
The primary aim of this study is to compare wound outcomes between two closure strategies after open appendectomy:

1. Simple interrupted skin sutures (standard method), versus
2. Subcuticular (intradermal) skin suture combined with a subcutaneous closed suction drain.

Specifically, the study aims to

* Determine whether the combined subcuticular closure with drain reduces the incidence of superficial surgical- site infection (SSI) within 30 days compared with interrupted sutures.
* Evaluate the effect of both techniques on secondary outcomes, including seroma or abscess formation, wound dehiscence, post-operative pain, cosmetic appearance of the scar, length of hospital stay, and drain-related adverse events.

DETAILED DESCRIPTION:
Open appendectomy remains a common emergency operation worldwide, particularly in settings where laparoscopic surgery is not feasible. Post-operative wound complications - especially superficial surgical-site infection (SSI), seroma and dehiscence - are frequent and lead to pain, longer hospital stay, antibiotic use and higher costs.

Reported SSI rates after appendectomy vary, but pooled global data suggest about 7 infections per 100 appendectomies, with higher rates generally seen after open procedures compared to laparoscopic approaches.

Skin closure technique is one modifiable factor influencing wound outcomes. Simple interrupted non-absorbable sutures are widely used, but continuous intradermal (subcuticular) absorbable sutures are increasingly studied. Randomized trials and systematic reviews show that subcuticular closure is at least as safe as interrupted closure regarding SSI, while often offering advantages such as improved cosmetic results, reduced need for suture removal, and lower patient discomfort.

A notable randomized trial in open appendectomy found fewer wound complications and better patient-reported outcomes with intradermal closure, though evidence across studies remains heterogeneous.

Placement of a subcutaneous closed suction drain is another potential strategy to reduce dead space and fluid collections, thereby lowering risks of seroma and infection. Meta-analyses suggest possible reductions in SSI and length of stay in abdominal surgery, but results are inconsistent and routine use remains controversial.

Current WHO guidelines on SSI prevention do not recommend a universal closure technique or routine subcutaneous drains, highlighting the need for targeted evidence.

Thus, the comparative effectiveness of simple interrupted sutures versus subcuticular closure combined with a subcutaneous drain in open appendectomy remains unclear, justifying a randomized controlled trial to address this gap.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years (or per local ethics), undergoing open appendectomy for acute appendicitis (elective not included).
* Skin incision for open appendectomy (McBurney/Gridiron or Lanz).
* Patient (or legal guardian) able and willing to provide informed consent.

Exclusion Criteria:

* Laparoscopic appendectomy or conversion to laparoscopic approach.
* Previous abdominal surgery at the same site (risk of altered wound healing).
* Pre-existing skin infection at the surgical site.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of superficial surgical-site infection (SSI) | 30 days
  Incidence of superficial surgical-site infection (SSI) after open appendectomy, defined according to CDC/NHSN criteria (purulent drainage, positive culture, or surgeon diagnosis).

SECONDARY OUTCOMES:
Incidence of other wound-related complications | 30 days
  * Seroma or subcutaneous abscess formation.
  * Wound dehiscence (partial or complete).
  * Drain-site infection or complications
Postoperative pain | at 24 hours, 48 hours, and 7-10days
  measured using the Visual Analogue Scale (VAS, 0-10 cm)

REFERENCES:
- [Result] Danwang C, Bigna JJ, Tochie JN, Mbonda A, Mbanga CM, Nzalie RNT, Guifo ML, Essomba A. Global incidence of surgical site infection after appendectomy: a systematic review and meta-analysis. BMJ Open. 2020 Feb 18;10(2):e034266. doi: 10.1136/bmjopen-2019-034266. PMID 32075838
- [Result] Allegranzi B, Bischoff P, de Jonge S, Kubilay NZ, Zayed B, Gomes SM, Abbas M, Atema JJ, Gans S, van Rijen M, Boermeester MA, Egger M, Kluytmans J, Pittet D, Solomkin JS; WHO Guidelines Development Group. New WHO recommendations on preoperative measures for surgical site infection prevention: an evidence-based global perspective. Lancet Infect Dis. 2016 Dec;16(12):e276-e287. doi: 10.1016/S1473-3099(16)30398-X. Epub 2016 Nov 2. PMID 27816413
- [Result] Ishinuki T, Shinkawa H, Kouzu K, Shinji S, Goda E, Ohyanagi T, Kobayashi M, Kobayashi M, Suzuki K, Kitagawa Y, Yamashita C, Mohri Y, Shimizu J, Uchino M, Haji S, Yoshida M, Ohge H, Mayumi T, Mizuguchi T. Recent evidence for subcutaneous drains to prevent surgical site infections after abdominal surgery: A systematic review and meta-analysis. World J Gastrointest Surg. 2023 Dec 27;15(12):2879-2889. doi: 10.4240/wjgs.v15.i12.2879. PMID 38222020
- [Result] Andrade LA, Munoz FY, Baez MV, Collazos SS, de Los Angeles Martinez Ferretiz M, Ruiz B, Montes O, Woolf S, Noriega JG, Aparicio UM, Gonzalez IG. Appendectomy Skin Closure Technique, Randomized Controlled Trial: Changing Paradigms (ASC). World J Surg. 2016 Nov;40(11):2603-2610. doi: 10.1007/s00268-016-3607-x. PMID 27283187
- [Result] Imamura K, Adachi K, Sasaki R, Monma S, Shioiri S, Seyama Y, Miura M, Morikawa Y, Kaneko T. Randomized Comparison of Subcuticular Sutures Versus Staples for Skin Closure After Open Abdominal Surgery: a Multicenter Open-Label Randomized Controlled Trial. J Gastrointest Surg. 2016 Dec;20(12):2083-2092. doi: 10.1007/s11605-016-3283-z. Epub 2016 Oct 3. PMID 27699563
- [Result] Bhangu A, Soreide K, Di Saverio S, Assarsson JH, Drake FT. Acute appendicitis: modern understanding of pathogenesis, diagnosis, and management. Lancet. 2015 Sep 26;386(10000):1278-1287. doi: 10.1016/S0140-6736(15)00275-5. PMID 26460662